CLINICAL TRIAL: NCT03097172
Title: The Effect of GRAVITY on Physiological Measurements During Invasive Coronary Angiography and Intervention
Acronym: GRAVITY
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Other Study IDs: B905
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention (PCI); Chronic Total Occlusion (CTO); Cardiac MRI; Fractional Flow Reserve (FFR); Doppler Flow Velocity; Cardiovascular Disease; Atherosclerosis; Hydrostatic Pressure
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Stable elective patients Stenotic coronary artery 10 x LAD 10 x RCA 10 x Cx
  30 patients total
- Group 2: Stable elective patients Chronic total occlusion of one artery
  10 x LAD 10 x RCA
  20 patients total

SUMMARY:
This is a single centre observational study on the impact of change in patient position and hence gravity, on physiological measurements in coronary arteries.

When patients present with heart attacks involving completely occluded heart arteries, there are signs anecdotally and in literature that arteries sitting higher up with the patient lying flat, receive less blood supply than arteries sitting lower down.

The investigators believe this effect is due to the pull of gravity on the flow of blood through the heart arteries. If this is indeed the case, changing position from lying supine (patient on their back) to lying prone (patient on their front) could reverse these anatomical positions and change measurements obtained during a coronary angiogram. These measurements include pressure and flow.

DETAILED DESCRIPTION:
The study will contain two groups:

Group 1 - stable elective patients with stenotic coronary arteries. These patients are referred as outpatients for a 'pressure wire' test.

Group 2 - stable elective patients with a chronic total occlusion of an artery (CTO). The artery will be either the left anterior descending artery (LAD) or right coronary artery (RCA)

Group 1 - 30 patients

Patients will be recruited from referrals to the centre for a pressure wire study. Participants will be screened for eligibility using the protocol inclusion and exclusion criteria. Study information will be given and informed consent obtained.

Patients will start the procedure prone. A physiology wire will be placed in the artery of interest and measurements taken. Patients will then be turned into the standard supine position with repeat measurements. The study is now completed. The usual pressure measurements will be taken and used to guide treatment as per standard protocol.

Group 2 - 20 patients

Patients will be recruited from referrals to the centre for a percutaneous coronary intervention (PCI) to a chronic total occlusion (CTO). Participants will be screened for eligibility using the protocol inclusion and exclusion criteria. Study information will be given and informed consent obtained.

Patients will undergo CTO PCI as per standard procedure. Once completed, the vessel will be occluded using balloon inflation. Physiological measurements will be taken distal to the occluded balloon. The patient will then be turned prone and repeat measurements again with balloon occlusion will be taken.

This group will have MRI scanning as part of standard care before the procedure. The study will carry out a further MRI, this time in the prone position before PCI as part of the study protocol

ELIGIBILITY:
Group 1

Inclusion Criteria:

1. Age > 18 years of age
2. Angina symptoms or evidence of myocardial ischaemia
3. Stenosis >50% in LAD or RCA on coronary angiogram or CT coronary angiogram
4. Participant is willing and able to give informed consent
5. Eligible for PCI

Exclusion Criteria:

1. Previous CABG with any patent grafts
2. Significant left main stem stenosis
3. Lesion of interest in Circumflex artery
4. Haemodynamic Instability
5. Unable to consent
6. Unable to receive dual antiplatelet therapy
7. Contraindication to adenosine
8. Recent acute coronary syndrome (ACS) (<48 hours)
9. Pregnancy
10. Unable to lie prone
11. Severe valvular heart disease or cardiomyopathy

Group 2

Inclusion Criteria:

1. Age >18 years of age
2. Stable angina / ischaemic symptoms / and / or
3. Evidence of viability and /or ischaemia in the chronic total occlusion (CTO) territory
4. Participant is willing and able to give informed consent.
5. Presence of chronic total occlusion (CTO) in LAD or RCA
6. Eligible for PCI to a chronic total occlusion (CTO)

Exclusion Criteria:

1. Previous CABG with any patent grafts
2. Significant left main stem stenosis
3. Dominant collateral supply from circumflex artery
4. Both LAD and RCA occluded
5. Haemodynamic instability
6. Unable to receive antiplatelet therapy
7. Contraindication to adenosine
8. Recent ACS (<48 hours)
9. eGFR<40
10. Pregnancy
11. Severe valvular heart disease or cardiomyopathy
12. Contraindication to Cardiac MRI
13. Unable to lie prone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the centre for 'pressure wire study' (group 1) or CTO PCI (group 2). Referred from secondary care to tertiary centre.
  Participants will be patients suffering from ischaemic heart disease living in the area served by the tertiary centre
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Coronary physiology changes | 5 minutes
  Changes in coronary physiology in the same vessel when comparing prone and supine patient position

SECONDARY OUTCOMES:
MRI finding | 4 weeks
  To observe any difference in ischaemia assessment when comparing prone and supine MRI

CONTACTS AND LOCATIONS:
Overall Officials: John R Davies, MBBS, PhD, Principal Investigator — Essex Cardiothoracic Centre, Basildon and Thurrock University Hospitals Foundation Trust
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No